CLINICAL TRIAL: NCT07342790
Title: Utilization of Artificial Intelligence in Supporting Physical Therapy Clinical Decision in Management of Myofascial Pain Syndrome Patients
Brief Title: Artificial Intelligence Clinical Decision
Acronym: AI/CDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Mohamed Abousaida, Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/006051
Record Dates: First submitted 2025-12-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Myofacial Pain Syndrome; Clinical Decision Support
Keywords: Clinical decision; artificial intelligence; pain; myofascial pain syndrome
MeSH Terms: conditions — Facial Neuralgia; Pain; Myofascial Pain Syndromes | interventions — Dry Needling; Muscle Stretching Exercises; Transcutaneous Electric Nerve Stimulation; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI.Group (Experimental): clinical decision making will depend on the integration of ChatGPT 4 into clinical decision-making process as a clinical advisor which recommends application of modalities based on clinical problems as follows dry needling for pain management, proprioceptive neuromuscular facilitation (PNF) stretching for muscle & joint rom enhancement, strengthening exercises (isometric & dynamic) for functional improvement and TENS (transcutaneous electrical nerve stimulation) in addition to home exercises as adjuvant therapies & ergonomic education
  Interventions: Procedure: dry needling; Other: neuromuscular facilitation (PNF) stretching; Other: strengthening exercises (isometric & dynamic); Device: Transcutaneous electrical nerve stimulation
- Traditional Group (Experimental): The traditional physical therapy treatment regime consists of hot pack (HP), transcutaneous electrical nerve stimulation (TENS), and ultrasound (US) for five days a week for two weeks, Application rules were:
  * Ultrasound (US): Continuous US at a frequency of 1 MHz was applied at a dose of 1.5 watt/cm² for six minutes daily.
  * Transcutaneous Electrical Nerve Stimulation (TENS): TENS was applied for 30 minutes daily.
  * Hot Pack (HP): HP was applied for 20 minutes daily.
  * In addition to these modalities, stretching exercises affected muscles
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Ultrasound; Other: Hot pack; Other: Stretching exercises

INTERVENTIONS:
Procedure: dry needling — Dry needling is a physical therapy intervention. It uses thin, solid filiform needles where no medication is injected, it targeting myofascial trigger points. The needle is inserted into the muscle tissue, and a local twitch response may occur which is considered a desired effect
  Arms: AI.Group
Other: neuromuscular facilitation (PNF) stretching — Proprioceptive neuromuscular facilitation stretching is a therapeutic stretching technique. It is commonly used in physical therapy and rehabilitation, involves stretching a target muscle , This is followed by an isometric or isotonic contraction
  Arms: AI.Group
Other: strengthening exercises (isometric & dynamic) — strengthening exercises are therapeutic interventions aiming to increase muscle strength and endurance. dynamic strengthening involves changes of the muscle length during contraction and isometric strengthening has no change of the muscle length
  Arms: AI.Group
Device: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation is a non-invasive modality which is commonly used for pain management through delivering low-voltage electrical currents that applied through surface electrodes on the skin.
Device: Ultrasound — Ultrasound is a therapeutic physical therapy modality which uses high frequency sound waves which are applied using coupling gel.
  Arms: Traditional Group
Other: Hot pack — Hot pack therapy is a superficial heat modality used in physical therapy, applied for a controlled duration, 20 minutes with A protective layer (towel) is placed between the pack and skin to prevent burns
  Arms: Traditional Group
Other: Stretching exercises — Stretching exercises are physical therapy interventions aimed at increasing muscle length and joint range of motion
  Arms: Traditional Group

SUMMARY:
The goal of this study is to investigate the effect of AI integration into clinical physical therapy clinical decision in improving cost effectiveness and clinical outcomes purposes of the study are:

1. Compare the effectiveness of AI driven and human driven clinical decision in physical therapy clinical practice on management of pain in myofascial pain syndrome.
2. Compare the effectiveness of AI driven and human driven clinical decision in physical therapy clinical practice on improving joint range of motion limitations in myofascial pain syndrome.
3. Compare the effectiveness of AI driven and human driven clinical decision in physical therapy clinical practice on improving muscle strength in myofascial pain syndrome.
4. Compare the effectiveness of AI driven and human driven clinical decision in physical therapy clinical practice on management of functional limitation in myofascial pain syndrome.
5. Compare the effectiveness of AI driven and human driven clinical decision in physical therapy clinical practice on cost-effectiveness in physical therapy management of myofascial pain syndrome.

DETAILED DESCRIPTION:
Evaluation of AI impact on health care processes still needs more investigation whatever the review of literature reveals, there is a great interest in developing AI tools to support clinical workflows, with increasing high-quality evidence being generated. Investigation of the impact of AI integration into the process of physical therapy clinical decision-making in management of myofascial pain syndrome still not examined or tested. The study planned to compare the efficacy using AI model to support physical therapy decision based on clinical problems solving by evaluating clinical outcomes such as pain intensity, muscular strength, joint rang motion, functional level and therapeutic cost effective compared to traditional clinical decision in patient with myofascial pain syndrome. Formulation A well-established detailed input (prompt) created to guide ChatGPT to what is requested and the proper way to process through the input to develop comprehensive, multimodal approaches (different modalities categories as therapeutic exercises, electrotherapy, complementary and manual approaches when indicated, evidence-based physiotherapy treatment protocol for and planning therapeutic interventions based on studies from PEDro, PubMed, Cochrane, Scopus, and Google Scholar. Patients will be assigned to two groups; one receives AI based clinical decision therapeutic interventions compared to the other group which will receive a traditional intervention according to published methods. Outcomes measures will be assed to compare which is more effective and result in best outcomes and less cost. Trail expected to test if it's valuable to use AI module in data analysis to support choice effective intervention and test the concept based on patient clinical problem-solving approach in physical practice against previously tested traditional methods, additional benefits may provide an assessment of a trail to formulate successful prompt to be used in other conditions. Although there are many studies in supporting clinical decision, still there are many questions concerned with the validity , methods , efficacy , cost effectiveness , scope and ethics of application

ELIGIBILITY:
Inclusion Criteria:

* A- Demographic: Adult individuals 18-65 both sex

B- Pain Characteristics:

* Localized pain.
* Intensity: baseline pain score of 4 or higher on the VAS . C- Duration: chronic pain 3-6 months

D- Prescence of Myofascial Trigger Points (MTrPs):

E- Daily Functioning limitations: moderate or severe

Exclusion Criteria:

* • Severe cognitive impairment or illness.

  * Recent history of major surgery or trauma (within 3 months).
  * Other chronic conditions that could significantly interfere with the study.
  * Patients with fibromyalgia which may have the Key Diagnostic Criteria for Fibromyalgia Syndrome:

    1. Widespread Pain Index (WPI) (appendix (2): Measures the number of painful areas across the body. A score of 7 or more indicates a higher likelihood of FMS (Wang et al. ,2025).
    2. Symptom Severity Scale (SSS) (appendix3): Assesses the severity of symptoms such as fatigue, sleep disturbances, and cognitive difficulties. A score of 5 or more is indicative of FMS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity changing | AI Group:12 sessions (1 every 3 days) Measures: Pre-1st, 4th,7th, 10th & post-12th session. Traditional Group:10 sessions/2weeks (5 daily, 2 days off, 5 daily)Measures: Pre-1st,4th,7th,10th & 2 days post-10th session
  Pain intensity is a subjective measurement of pain level or magnitude that can be Measured using a visual analog scale (VAS) , which is a tool used for measuring intensity of pain. It consists of a 10-centimeter line with endpoints defining extremes of pain (e.g., "no pain" to "worst possible pain"). A quantitative indicator of pain intensity will be provided by participants marking their level of pain on the line.

SECONDARY OUTCOMES:
Functional level Assessment | AI Group:12 sessions (1 every 3 days) Measures: Pre-1st, 4th,7th, 10th & post-12th session. Traditional Group:10 sessions/2weeks (5 daily, 2 days off, 5 daily)Measures: Pre-1st,4th,7th,10th & 2 days post-10th session
  Functional level refers to a patient's ability to perform activities of daily living (ADLs) and special tasks which reflect overall physical capacity, independence, and quality of life. Patient-Specific Functional Scale (PSFS) allows participants to identify and rate specific activities that they find difficult due to their pain. They rate their ability to perform these activities on a scale from 0 (unable to perform) to 10 (able to perform at prior level). This instrument will evaluate functional improvement in daily living activities, customized to the unique limitations of each participant, offering a customized assessment of therapeutic success.
Assessment of Joint Range Motion changes | AI Group:12 sessions (1 every 3 days) Measures: Pre-1st, 4th,7th, 10th & post-12th session. Traditional Group:10 sessions/2weeks (5 daily, 2 days off, 5 daily)Measures: Pre-1st,4th,7th,10th & 2 days post-10th session
  The joint ROM refers to the extent of movement at a joint necessary to displace a bone within its spatial limits, Using Digital goniometer is an instrument used to measure and assessment of joint angles of the human body, in biomechanics, rehabilitation, and clinical research. Digital Goniometer is a new version alternative to the traditional mechanical goniometer that provides precise digital reading for angle measurement.

CONTACTS AND LOCATIONS:
Overall Officials: HESHAM M ABOUSAIDA, master, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic, faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No